CLINICAL TRIAL: NCT01051635
Title: A Phase I Study of Indenoisoquinolines LMP400 and LMP776 in Adults With Relapsed Solid Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100056; 10-C-0056; NCT01245192 (obsolete NCT alias)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Neoplasms; Lymphoma
Keywords: DNA Repair; DNA Damage; Advanced Cancer; Advanced Malignancies; Topoisomerase Inhibitor
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — NSC 724998; indimitecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): LMP400 administered IV daily for 5 days per dose escalation table.
  Interventions: Drug: LMP400
- Cohort B (Experimental): LMP776 administered IV daily for 5 days per dose escalation table.
  Interventions: Drug: LMP776

INTERVENTIONS:
Drug: LMP400 — Indenoisoquinolines are non-camptothecin inhibitors of topoisomerase 1 with improved characteristics such as better chemical stability, producing stable DNA-top1 cleavage complexes, and exhibiting a preference for unique DNA cleavage sites compared with their camptothecin counterparts.
  Arms: Cohort A
Drug: LMP776 — Indenoisoquinolines are non-camptothecin inhibitors of topoisomerase 1 with improved characteristics such as better chemical stability, producing stable DNA-top1 cleavage complexes, and exhibiting a preference for unique DNA cleavage sites compared with their camptothecin counterparts.
  Arms: Cohort B

SUMMARY:
Background:

* Indenoisoquinolines are experimental cancer treatment drugs that damage the DNA in cells, resulting in cell death. Researchers have been studying these drugs and their usefulness in treating types of cancer that have not responded well to standard therapies like surgery or radiation.
* LMP400 (NSC 743400) and LMP776 (NSC 725776) are indenoisoquinolines that have not been given to cancer patients before. These drugs have very similar chemical structures and work the same way, but researchers do not know which one will work best. More information is needed about how LMP400 and LMP776 are processed by the body and how effective they are in treating difficult-to-treat types of cancer.

Objectives:

* To determine the maximum tolerated dose of LMP400 (NSC 743400) and LMP776 (NSC 725776).
* To study how the body handles LMP400 and LMP776.
* To evaluate the effectiveness of LMP400 and LMP776 as a treatment for tumors and lymphoma that have not responded to standard treatment.

Eligibility:

- Individuals at least 18 years of age who have malignant solid tumors or Hodgkin s disease/non-Hodgkin lymphoma that has not responded to standard therapies.

Design:

* Participants will receive either LMP400 or LMP776. The treatment cycle will be 28 days. On the first 5 days of each cycle, participants will receive intravenous doses of their specific study drug, followed by 23 days without the drug. The 28-day cycle will be repeated as long as the drug does not cause severe side effects and the cancer remains stable or improves. The study doctor may increase or decrease the dose of study drug depending on how well it is tolerated.
* Blood, urine, and hair samples and skin and tumor biopsies will be collected during the first treatment cycle. Routine blood samples will be taken throughout the study.
* Other tests, including additional blood and urine samples, computed tomography (CT) or other scans, and bone marrow samples, may be performed as directed by the study doctors.

DETAILED DESCRIPTION:
Background:

* Indenoisoquinolines are non-camptothecin inhibitors of topoisomerase 1 (top1) with improved characteristics over their predecessors. Indenoisoquinolines have better chemical stability, producing stable DNA-top1 cleavage complexes, and exhibit a preference for unique DNA cleavage sites, compared with their camptothecin counterparts.
* They have demonstrated activity against camptothecin-resistant cell lines and produce DNA-protein crosslinks, which are resistant to reversal. They also show less or no resistance to cells overexpressing the ATP-binding cassette (ABC) transporters, ABCG2, and multidrug resistance (MDR-1).

Primary Objectives:

* Define the maximum tolerated dose (MTD) of LMP400 (NSC 743400) and LMP776 (NSC 725776) administered intravenously (IV) daily for 5 days (QDx5).
* Define the dose-limiting toxicities (DLTs) and toxicity profile associated with administration of LMP400 and LMP776.
* Evaluate the effect of LMP400 and LMP776 on the pharmacodynamic (PD) endpoint, gamma-H2AX, in tumor biopsy pre- and post-treatment. In particular, compare the PD response, defined as the mean percent nuclear area that is gamma-H2AX positive (%NAP) in tumor biopsies, at the MTD for LMP400 and LMP776, and the toxicity profile versus PD dose-response relationship.

Secondary Objectives:

* Obtain preliminary evidence of anti-tumor activity of LMP400 and LMP776.
* Characterize the pharmacokinetic (PK) profile of LMP400 and LMP776.

Eligibility:

-Adult patients must have histologically confirmed relapsed solid tumor malignancy or lymphoma that is metastatic or unresectable for which standard curative measures do not exist or are associated with minimal patient survival benefit.

Study Design:

* Cycle 1 and subsequent cycles: Patients will be randomized to receive either LMP400 or LMP776 administered IV QD over 1 hour on days 1-5 followed by 23 days without drug (28-day cycle).
* PK and PD samples will be collected in cycle 1 only. Tumor biopsies will not be collected during the escalation phase; however, tumor biopsies will be mandatory during the expansion phase.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically documented (confirmed at the Laboratory of Pathology, NCI), relapsed solid tumor malignancy or Hodgkin s disease/non-Hodgkin lymphoma that is metastatic or unresectable for which standard curative measures do not exist, or are associated with minimal patient survival benefit.
* Patients must have measurable or evaluable disease.
* Patients must have recovered to at least eligibility levels due to adverse events (AEs) and/or toxicity of prior chemotherapy or biologic therapy. They must not have had chemotherapy or biologic therapy within 4 weeks (6 weeks for nitrosoureas and mitomycin C, or 2 months for UCN-01), or therapy with tyrosine kinase inhibitors within 5 times the half-life of the inhibitors prior to entering the study. Patients must be (Bullet)2 weeks since any investigational agent administered as part of a Phase 0 study (also referred to as an early Phase I study or pre-Phase I study where a sub-therapeutic dose of drug is administered) at the PI s discretion, and should have recovered to eligibility levels from any toxicities.
* Patients must have recovered to at least a Grade less than or equal to toxicity eligibility levels due to adverse events (AEs) and/or toxicity of prior chemotherapy or biologic therapy. They must not have had chemotherapy or biologic therapy within 4 weeks (6 weeks for nitrosoureas and mitomycin C, or 2 months for UCN-01), or therapy with tyrosine kinase inhibitors within 5 times the half-life of the inhibitors prior to entering the study. Patients must be greater than or equal to 2 weeks since any prior administration of study drug in an exploratory IND/Phase 0 study. Patients must be greater than or equal to 1 month since completion of any prior radiation (greater than or equal to 2 weeks for palliative radiation therapy). However, patients receiving bisphosphonates for any cancer or undergoing androgen deprivation therapy for prostate cancer are eligible for this therapy. Prior therapy with topoisomerase I inhibitors is allowed.
* Age greater than or equal to 18 years.
* The Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
* Life expectancy greater than 3 months.
* Patients must have normal or adequate organ and marrow function as defined below:

  * Absolute neutrophil count greater than or equal to 1,500/microL
  * Platelets greater than or equal to 100,000/microL
  * Total bilirubin* within less than or equal to 1.5 normal institutional limits
  * AST (SGOT)/ALT (SGPT) less than or equal to 2.5 times institutional upper limit of normal
  * Creatinine less than 1.5 times upper limit of normal

OR

* Creatinine clearance greater than or equal to 60 mL/minute for patients with (measured) creatinine levels greater than or equal to 1.5 times upper limit of normal

  *we will allow patients with Gilbert s syndrome with total bilirubin up to 2.5 mg/dL
  * The effects of indenoisoquinolines on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry, for the duration of study participation, and for 2 months after discontinuation from the study. Women of child bearing potential must have a negative pregnancy test in order to be eligible. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Because there is an unknown but potential risk to nursing infants secondary to treatment of the mother with indenoisoquinolines, breastfeeding should be discontinued if the mother is treated with indenoisoquinolines.
  * Willingness to undergo skin biopsies.
  * At the point when tumor biopsies become mandatory rather than optional, disease amenable to biopsy and willingness to undergo biopsies or patient will be undergoing a procedure due to medical necessity during which the tissue may be collected, or tumor biopsy tissue from a previous research study or medical care is available for submission at registration. Criteria for the submission of tissue are:
* Tissue must have been collected within 3 months prior to registration
* Patient has not received any intervening therapy for their cancer since the collection of the tumor sample
* Tumor tissue must meet the minimum requirements outlined in Section 9.1.

  * Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients receiving any other investigational agents.
* Patients with known brain metastases are excluded from this clinical trial, with the exception of patients whose brain metastatic disease status has remained stable for greater than or equal to 2 months after treatment of the brain metastases, without steroids or anti-seizure medications. These patients may be enrolled at the discretion of the principal investigator.
* Patients with clinically significant illnesses which could compromise participation in the study, including, but not limited to, active or uncontrolled infection, immune deficiencies, known HIV infection requiring antiretroviral therapy, Hepatitis B, Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-01-25 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Safety | 1 cycle (28 days)
  Defined dose-limiting toxicities and toxicity profile associated with administration of LMP400 and LMP776

SECONDARY OUTCOMES:
Pharmacodynamic effects | Cycle 1 Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] O'Sullivan Coyne G, Kummar S, Rubinstein LV, Wilsker D, Moore N, Hogu M, Piekarz R, Covey J, Beumer JH, Ferry-Galow KV, Villaruz LC, Hollingshead MG, Holleran JL, Deppas JJ, Pommier Y, Ko B, Johnson BC, Parchhment RE, Ivy P, Doroshow JH, Chen AP. Phase 1 studies of the indenoisoquinolines LMP776 and LMP744 in patients with solid tumors and lymphomas. Cancer Chemother Pharmacol. 2025 May 29;95(1):58. doi: 10.1007/s00280-025-04778-5. PMID 40439882
- [Derived] Beumer JH, Kennard BC, Holleran JL, Moore N, Zlott J, Miller BM, Kummar S, Chen A, Doroshow J, Park W, Gobburu J, Dunn A. Evaluating the indotecan-neutropenia relationship in patients with solid tumors by population pharmacokinetic modeling and sigmoidal Emax regressions. Cancer Chemother Pharmacol. 2023 Mar;91(3):219-230. doi: 10.1007/s00280-023-04509-8. Epub 2023 Feb 23. PMID 36813886
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0056.html